CLINICAL TRIAL: NCT00094848
Title: A Multi-Center, Open-Label, Dose-Escalation Study to Evaluate the Safety, Efficacy, and Exposure to TRM-1 (Fully Human Monoclonal Antibody to the TRAIL-R1) in Subjects With Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Study of TRM-1 (TRAIL-R1 Monoclonal Antibody) in Subjects With Relapsed or Refractory Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRM1-HM01
Record Dates: First submitted 2004-10-27; First posted 2004-10-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — mapatumumab

INTERVENTIONS:
Drug: TRAIL-R1 mAb (TRM-1; HGS-ETR1)

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and exposure to TRM-1 in subjects with relapsed or refractory Non-Hodgkin's Lymphoma (NHL).

ELIGIBILITY:
Primary Inclusion Criteria:

* Relapsed or refractory histologically confirmed Non-Hodgkin's Lymphoma
* Previously treated with at least 1 therapeutic regimen and relapsed or progressed or failed to achieve a response after the last regimen
* 18 years of age or older

Primary Exclusion Criteria:

* Received a non-FDA approved investigational agent within the last 4 weeks
* Received cancer therapies (chemotherapy, biological therapy [including hormonotherapy], radiation therapy or immunosuppressants within the last 3 weeks, 8 weeks for monoclonal antibodies, radioimmunotherapy or nitrosourea
* Eligible for a hematopoietic stem cell transplant (HSCT) or have had an autologous HSCT within the last 16 weeks
* Prior history of an allogeneic HSCT
* HIV, AIDS-related lymphoma, central nervous system (CNS) lymphoma, Hepatitis-B or Hepatitis-C
* Infection requiring antibiotics within the last 4 weeks
* Major surgery within the last 4 weeks
* Pregnant or breast-feeding women
* History of other cancers within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Primary Completion 2006-12 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas